CLINICAL TRIAL: NCT02149446
Title: Pancreas Fistula After Distal Pancreatic Resection: Prevention and Treatment in a Randomized Controlled Trial
Brief Title: Does Reinforcement of the Staple Line in Left Pancreatectomy Reduce the Rate of Pancreatic Fistula?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other); Lund University Hospital (Other); University Hospital, Linkoeping (Other); Norrlands University Hospital (Other)
Responsible Party: Principal Investigator, John Blomberg, MD PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Surgisis-001
Record Dates: First submitted 2014-05-21; First posted 2014-05-29 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Post Operative Pancreatic Fistula
Keywords: Left sided pancreatic resections; Distal pancreatic resections; Reinforced staple line; Post operative pancreatic fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgisis reinforcement of staple line (Experimental): The stapler used to divide the pancreas is reinforced with Surgisis (COOK Medical).
  Interventions: Device: Surgisis (C-SLRA-ECH60) made by COOK Medical
- No reinforcement of staple line (No Intervention): The stapler used to divide the pancreas is not reinforced with any material

INTERVENTIONS:
Device: Surgisis (C-SLRA-ECH60) made by COOK Medical — Surgisis is extracellular matrix collagen made of the submucosal layer of pigs intestines. Surgisis is gradually remodeled, leaving behind organized tissue
  Other Names: Surgisis reinforcement of staple line
  Arms: Surgisis reinforcement of staple line

SUMMARY:
Dividing pancreas when performing left-sided resections opens the risk for leakage from the divided end of the pancreas. Pancreatic juices could have a severe effect on surrounding abdominal tissues with abscess formation producing systemic inflammation and potential lethal bleeding.

Studies have shown that reinforcement of the staple line when dividing pancreas could reduce the risk of leakage.

Surgisis (COOK Medical) a product already in use for staple line reinforcement in gastric and lung surgery could be used as a reinforcement when stapling pancreas in left sided resections.

In a prospective randomized trial we want to compare Surgisis reinforcement to no reinforcement of stapled division in left sided pancreatic resections.

Primary outcome is pancreatic fistula yes/no.

DETAILED DESCRIPTION:
Resection of the distal pancreas is often done due to a localized tumor in the body or tail of the pancreas. During later years the mortality after pancreatic resections have been reduced but there still is a substantial risk of severe complications mainly due to leakage from the pancreatic division line which could lead to suffering, longer hospital stay, higher costs and sometimes death. Leakage from a tail resection is probably more common than thought of before. Frequencies of above 30% and even up to 60% have been reported.

The use of somatostatin to reduce the production of pancreatic juice or comparison between stapled division, suturing of the remaining part of the cut pancreas or covering it with glue or available surrounding tissue have not showed significant superiority for any of these methods except for a positive trend regarding the stapling technique. Staple line reinforcement with resorbable mesh has in some studies showed a both negative and positive effect on pancreatic fistula frequency. These studies have been small and non-randomized. A larger randomized single blinded study by Hamilton et al on the other hand showed a significant positive effect on pancreatic fistula frequency after distal pancreatic resection using an absorbable reinforcement device put on the stapler, when only regarding type B and C fistulas as defined by the ISGPF (International Study Group on Pancreatic Fistula) pancreatic leak grading system.

Although all these endeavors the problem of pancreatic fistulas remain and therefore all these operations are concluded with the deposit of one or more drains to the area of the cut pancreas.

There is therefore of importance to continue the work of reducing complications in high risk pancreatic surgery using scientific procedures of high quality as in blinded randomized controlled trials (RCT). The use of reinforced stapling techniques has been used in lung surgery and bariatric surgery to reduce air leakage and strengthen anastomoses. The material used is processed submucosa from the small bowel of the pig, produced by COOK© Medical to fit endoscopic staplers from Ethicon© or Covidien©.

After the promising result from Hamilton et al we plan to study if the reinforcement made by COOK© could reduce the frequency of pancreatic fistula after stapled distal pancreatic surgery in a single blinded RCT.

ELIGIBILITY:
Inclusion Criteria:

* Every patient eligible for pancreatic tail resection.

Exclusion Criteria:

* Not able to read Swedish.
* Not able to understand or accept the concept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Post operative pancreatic fistula (POPF), Y/N | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Pancreatic amylase concentration in any post operative drains. Fistula is diagnosed if pancreatic amylase > 3 times the upper normal limit of pancreatic amylase in plasma on post operative day 3 or later

SECONDARY OUTCOMES:
POPF healing time | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Time from diagnosis to healed pancreatic fistula
POPF grade according to International Study Group of Pancreatic Fistula (ISGPF) grade A/B/C | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Worst POPF grade registered during the observation period.
Blood chemistry | The first 7 days after operation
  During the first 7 post operative days each participant will have daily measurements taken from blood samples regarding C-reactive protein, white blood count, pancreatic plasma amylase and from drain fluid regarding pancreas amylase. The participants daily drain volume will also be measured.
Morbidity | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
  According to Clavien scoring
Mortality | < 90 days after the operation
Hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
  Number of days

CONTACTS AND LOCATIONS:
Overall Officials: John Blomberg, MD, PhD, Principal Investigator — Dep of Surgical Gastoenterology, Karolinska University Hospital, Stockholm, Sweden
Locations (1):
- Dep of Surgical Gastroenterology, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Wennerblom J, Ateeb Z, Jonsson C, Bjornsson B, Tingstedt B, Williamsson C, Sandstrom P, Ansorge C, Blomberg J, Del Chiaro M. Reinforced versus standard stapler transection on postoperative pancreatic fistula in distal pancreatectomy: multicentre randomized clinical trial. Br J Surg. 2021 Apr 5;108(3):265-270. doi: 10.1093/bjs/znaa113. PMID 33793753